CLINICAL TRIAL: NCT01597115
Title: ENhancing Maturation of Autogenous Arteriovenous Hemodialysis Access by Aggressive surveillaNCe With Duplex and Endovascular Treatment
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUPLEX-IV-02-12
Record Dates: First submitted 2012-05-10; First posted 2012-05-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2014-05

CONDITIONS: End Stage Renal Disease
Keywords: duplex study; hemodialysis access; maturation rate; endovascular intervention
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duplex (Active Comparator): Patients in this group will be examed by duplex ultrasonography at 2 and 4 weeks after surgery
  Interventions: Procedure: Duplex ultrasonography
- physical exam (No Intervention): According to the K/DOQI guideline, patients will be examed by vascular access surgeon at 2 and 4 weeks after surgery

INTERVENTIONS:
Procedure: Duplex ultrasonography
  Arms: Duplex

SUMMARY:
The aim of this study is to evaluate whether Aggressive duplex surveillance after vascular access surgery with native vein for hemodialysis can increase the maturation rate of arteriovenous fistula. This study will be conducted as a single center, prospective, 1:1 randomized study. Enrolled patients will be randomized as a control group (Physical exam at 2 and 4 weeks after surgery) and duplex group (duplex study and physical exam at 2 and 4 weeks after surgery). Maturation of arteriovenous fistula will be evaluated at 8 weeks after surgery by duplex in all patients.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal disease
* newly formed hemodialysis access with native vein
* 20~70 years

Exclusion Criteria:

* hemodialysis access surgery with ePTFE graft
* hemodialysis access surgery with basilic vein transposition
* hemodialysis access surgery with brachial vein transposition
* cephalic vein < 2.5mm in diameter
* radial artery diameter <2.0mm in radiocephalic arteriovenous fistula

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
hemodialysis access maturation rate | 8 weeks after surgery

SECONDARY OUTCOMES:
factors predicting maturation failure | 8 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Il Min, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea